CLINICAL TRIAL: NCT03487601
Title: Transcranial Direct Current Stimulation (tDCS) to Improve Fatigue and Cognitive Function During Breast Cancer Chemotherapy: A Feasibility Study
Brief Title: Transcranial Direct Current Stimulation (tDCS) to Improve Fatigue and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Robert L. Sloan Fund for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: J17138; IRB00140819 (Other: JHMIRB)
Record Dates: First submitted 2018-02-02; First posted 2018-04-04 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer; Fatigue
Keywords: docetaxel; Stage I - IV; chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The proposed feasibility trial is a randomized, sham-controlled, double-blind experiment.
Who Masked: Participant
Masking Description: Participants will be randomized to either active or sham tDCS and will undergo 5 consecutive treatments of daily tDCS beginning the Monday following the first day of their on-study chemotherapy cycle. Active treatment will consist of a mild electrical current (2mA) administered via saline-soaked sponge electrodes placed along the intact scalp for 30 minutes a day for five days. Sham stimulation will involve brief delivery of current in a manner that does not result in changes in neuronal firing patterns, but that is perceived as active treatment by participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Active transcranial direct current stimulation: Participants will undergo five consecutive days (Monday-Friday) of active stimulation beginning the Monday after their on-study chemotherapy administration. Questionnaires and cognitive assessment will be completed on the first and last days of stimulation (i.e., Monday and Friday). On all 5 days, participants will engage in cognitive tasks while receiving stimulation (either active or sham) in order to maximize stimulation effects 43. In order to assess for duration of subjective effects, participants will complete self-report measures of subjective fatigue, cognitive function and QOL immediately prior to their next chemotherapy (approximately 10-14 days after completion of stimulation).
  Interventions: Other: transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Sham transcranial direct current stimulation: Participants will undergo five consecutive days (Monday-Friday) of sham stimulation beginning the Monday after their on-study chemotherapy administration. Questionnaires and cognitive assessment will be completed on the first and last days of stimulation (i.e., Monday and Friday). On all 5 days, participants will engage in cognitive tasks while receiving stimulation (either active or sham) in order to maximize stimulation effects 43. In order to assess for duration of subjective effects, participants will complete self-report measures of subjective fatigue, cognitive function and QOL immediately prior to their next chemotherapy (approximately 10-14 days after completion of stimulation).
  Interventions: Other: sham transcranial direct current stimulation

INTERVENTIONS:
Other: transcranial direct current stimulation — Active treatment will consist of a mild electrical current (2mA) administered via saline-soaked sponge electrodes placed along the intact scalp for 30 minutes a day for five days.
  Other Names: tDCS
  Arms: Active tDCS
Other: sham transcranial direct current stimulation — Sham stimulation will involve brief delivery of current in a manner that does not result in changes in neuronal firing patterns, but that is perceived as active treatment by participants.
  Other Names: sham stimulation
  Arms: Sham tDCS

SUMMARY:
This research is being done to determine whether transcranial direct current stimulation (tDCS) can improve fatigue and certain thinking skills in women with breast cancer receiving chemotherapy.

Transcranial Direct Current Stimulation is a form of brain stimulation during which low amounts of electrical current are delivered to the brain using electrodes attached to the scalp. The idea of using electrical stimulation to affect neurological symptoms has been around for more than 100 years with the first reported use in 1801. Since the 1960s, tDCS has been used in research for a variety of reasons including stroke rehabilitation, memory enhancement and for depression.

People aged 18 or older who are currently receiving chemotherapy with docetaxel and who are experiencing fatigue may join.

DETAILED DESCRIPTION:
Fatigue and cognitive impairment are commonly reported symptoms associated with impaired quality of life (QOL) and productivity in breast cancer patients receiving chemotherapy. Working memory, the brain's system for temporarily storing and manipulating information required to carry out more complex cognitive tasks, is particularly affected by cancer and its treatment.

In women who have undergone chemotherapy for breast cancer, neuroimaging studies show structural brain changes as well as functional inefficiencies in a region critical for working memory, the left dorsolateral prefrontal cortex (DLPFC). Fatigue appears to play a critical role in the recruitment of the DLPFC during cognitive tasks.

Transcranial direct current stimulation (tDCS) is a safe, portable, non-invasive form of electrical brain stimulation that enhances neuronal transmission beneath scalp electrodes. Our group and others have shown that when applied to the left DLPFC, tDCS improves energy in patients with fatiguing medical conditions and that it improves cognition in both healthy adults and those with neurodegenerative diseases.

The proposed feasibility trial is a randomized, sham-controlled, double-blind experiment. Eligible individuals will be ≥ age 18 years with stage I-IV breast cancer undergoing docetaxel-based chemotherapy every 3 weeks (at least 60 mg/m2 dose) with or without HER2-targeted therapy who self-report moderate or severe fatigue (rated ≥ 4 on a scale of 0-10) during at least 3 days of their most recent chemotherapy cycle. Participants will be randomized to either active or sham tDCS and will undergo 5 consecutive treatments of daily tDCS beginning the Monday following the first day of their on-study chemotherapy cycle. Active treatment will consist of a mild electrical current (2mA) administered via saline-soaked sponge electrodes placed along the intact scalp for 30 minutes a day for five days. Sham stimulation will involve brief delivery of current in a manner that does not result in changes in neuronal firing patterns, but that is perceived as active treatment by participants.

Participants will complete self-report measures of fatigue, cognitive function and QOL along with cognitive testing at the beginning and end of the five-day intervention. Subjective fatigue, QOL and cognitive function will be also assessed prior to administration of the next cycle of chemotherapy. Total time on study will be approximately 3 weeks (one cycle of chemotherapy). Daily subjective fatigue will be monitored throughout participation.

ELIGIBILITY:
Inclusion Criteria:

* Women or men, 18 years of age or older
* Stage I-IV breast cancer receiving docetaxel-based chemotherapy (at least 60 mg/m2) every 21 days

  • Docetaxel may be administered concurrently with other chemotherapy agents and/or with HER2 targeted therapies at the discretion of the treating provider
* Fatigue: Self-report of moderate or severe fatigue on at least 3 days during the prior cycle of docetaxel-based chemotherapy, defined as ≥ 4 on a 0 (no fatigue) to 10 (worst fatigue imaginable) scale.
* Able and willing to complete study tasks as evidenced by at least the following according to the assessment of a study team member: fluent English speaker; hearing and language comprehension; and, sufficient literacy to complete study forms and questionnaires
* Patient understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form.

Exclusion Criteria:

* Dementia as assessed by a MMSE score < 24 on initial screening.
* Known pregnancy or nursing.
* Any of the following: known diagnosis of schizophrenia or bipolar disorder, seizure disorder, pacemaker, hearing aids, any metal implanted in the head, untreated hypothyroidism, aphasia, delirium, known neurologic disorder which affects cognitive function, prior traumatic brain injury, known heart failure

  • Note: presence of a mediport is not an exclusion criteria
* Use of the following medications for seven days prior to and during study participation:

  * Stimulant medications
  * Carbamazepine/Tegretol
  * Cough/cold medicines (e.g. Dextromethorphan, Triaminic, Robitussin, Vics Formula 44)
  * Flunarizine/Sibelium
  * Propanolol/Inderal
  * Sulpiride
  * Pergolide
  * Rivastigmine/Exelon
  * Carbidopa/levodopa or levodopa
  * Ropinirole/Requip
  * Nicotine patch
* Use of illicit drugs for seven days prior to and during study participation.
* Self-reported consumption of > 14 alcoholic drinks per week or positive screening on the CAGE questionnaire in relation to the past year. NOTE: A single, standard alcoholic drink is defined as 10 grams of alcohol, which is equivalent to 285 mL of beer, 530 mL of light beer, 100 mL of wine or 30 mL of liquor.
* Skin conditions involving open sores on the scalp that would prevent proper application of the electrodes.
* Hairstyles that obstruct placement of the electrodes including cornrows, dreadlocks, braids or other hair accessories that cannot be removed.
* Known history of brain metastases or leptomeningeal carcinomatosis (even if adequately treated)
* Prior brain surgery
* Other medical or other condition(s) that in the opinion of the investigators might compromise the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-02-16 (Actual); Study Completion 2019-02-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of tDCS | Day 5
  Evaluation of the feasibility of 5 consecutive days of tDCS in breast cancer patients receiving docetaxel-based chemotherapy. Feasibility will be evaluated by assessing the proportion of study participants who complete at least 4 of 5 days of the planned tDCS intervention (active or sham) during docetaxel-based chemotherapy. If >80% of participants complete 4 of the 5 planned stimulation sessions, tDCS will be defined as feasible.

SECONDARY OUTCOMES:
Fatigue | Day 1, Day 5, and at End of study (approximately 3 weeks)
  Participants will complete self-report measures of fatigue. The Multidimensional Fatigue Symptom Inventory 30-item Short Form (MFSI-SF) will serve as the primary measurement tool for the assessment of subjective fatigue. This questionnaire assesses participants' subjective ratings across five subscales: general fatigue, physical fatigue, emotional fatigue, mental fatigue, and vigor. Responses are provided on 5-point Likert-like scales addressing the extent to which each symptom was experienced during the preceding 7 days ranging from 0 (not at all) to 4 (extremely). The subscale scores are obtained by summing scores within each subscale. The MFSI-SF total score is obtained by subtracting the vigor subscale score from the sum of the four fatigue subscales. Scores range from -36 to 144. The MFSI-SF is well validated in breast cancer patients. Breast cancer patients with fatigue produce an average score of 14.7 ± 15.2. The MFSI-SF takes approximately 5 minutes to complete.
Subjective Cognitive Function | Day 1, Day 5, and at end of study (approximately 3 weeks)
  Participants will self-report measures of cognitive function at the beginning and end of the five-day intervention. The endpoint for subjective cognition will be scores on the FACT-Cog, a 37-item self-report measure. Responses are provided on 5-point Likert-like scales addressing the frequency with which each type of cognitive difficulty occurred from 0 (never) to 4 (several times a day) over the prior seven days. Two additional subscales address "noticeability" or comments from others regarding cognition and "effect of perceived cognitive impairment on quality of life." These are rated on 5-point Likert-like scales ranging from 0 (not at all) to 4 (very much). The total FACT-Cog score is obtained by summing the individual subscale scores and ranges from 0 to 148. Breast cancer patients produce a mean FACT-Cog total score of 119.0 ± 23.3.The FACT-Cog takes approximately 5 minutes to complete.
Objective Cognitive Function | Day 1 and Day 5
  Objective cognitive function from baseline (prior to tDCS) to completion of tDCS will be assessed. The measurement tool for objective cognitive function for this objective will be the Paced Auditory Serial Addition Test (PASAT) of working memory. The PASAT is working memory task that has been well-validated medical populations including breast cancer. Test administration involves the aural presentation of single digits via computer in order to ensure a standardized rate of stimulus presentation. Stimuli are presented every three seconds (trial 1) or every two seconds (trial 2). Participants add each new digit to the one immediately prior as the test continues to present stimuli. The test score reflects the total number of correct sums given (out of 60 possible) in each trial. Two equivalent, alternative PASAT forms will be used to minimize practice effects. The test takes approximately 10 minutes to complete.
Quality of Life | Day 1, Day 5, End of study (approximately 3 weeks)
  The measurement tool for QOL will be the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). The impact of tDCS on QOL will be assessed by the EORTC QLQ-C30. This 30-item questionnaire includes five functional scales (physical, role, emotional, social and cognitive), three symptom scales (fatigue, nausea/vomiting and pain), a global health status scale and six single items (dyspnea, constipation, diarrhea, appetite, sleep and financial difficulty). The first 28 questions are answered using a Likert-like scale ranging from 1, "not at all", to 4, "very much". The last two questions are answered on a Likert-like scale ranging from 1, "poor" to 7, "excellent". The recall period is 7 days. The EORTC QLQ-C30 has been extensively used as a quality of life measure in breast cancer clinical trials and is well validated in the breast cancer population. The EORTC QLQ-C30 takes approximately 5 minutes to complete.

OTHER OUTCOMES:
Daily Fatigue | Daily from Day 1 to End of study (approximately 3 weeks)
  Daily subjective fatigue will be measured by the MD Anderson Brief Fatigue Inventory (BFI). The BFI will be completed daily from day 1 of stimulation until day 1 of the next chemotherapy cycle. Participants will be given multiple copies of the BFI with the date marked on them to complete at home. Participants will return the completed BFI at a follow-up visit or by mail. The BFI measures the severity of fatigue and the degree to which it interferes with function. The BFI has 9 items. The first 3 items rate fatigue severity and are measured on a scale of 0, "no fatigue", to 10, fatigue "as bad as you can imagine." The remaining items rate interference of fatigue and are measured on a scale of 0, "does not interfere" to 10, "completely interferes." The recall period for the BFI is 24 hours. The BFI has been validated in patients with solid tumors including breast cancer and in patients receiving chemotherapy. The BFI takes only a few minutes to complete.
Patient-Reported Side effects of tDCS | Before and after study intervention on Days 1, 2, 3, 4, 5
  Patient-Reported Side effects of tDCS will be assessed by a side effects questionnaire. This will include questions regarding physical sensations and mood experienced prior to and following each stimulation session (i.e. twice during all five sessions) to document the presence and severity of any tDCS-related side effects. Participants will be asked to rate the severity of these experiences and to report any other sensations they were not asked about directly. At the end of stimulation on the fifth day, each participant will also be asked whether he/she believes he/she was receiving active or sham tDCS as part of the side effects questionnaire and he/she will rate the degree of confidence with respect to these judgments. This questionnaire takes less than five minutes to complete.
Cognitive Function other than working memory (TMT) | Before and after study intervention on Days 1-5
  The measurement tool for objective cognitive function for this objective will be the Trail Making Test (TMT). The TMT is composed of 2 parts (A and B). Part A is designed to evaluate visual motor scanning and processing speed. Part B is designed to evaluate processing speed and executive functioning. These tests require patients to connect circles in numerical (part A) or alternating numerical and alphabetical sequence (part B) as quickly as possible. Results are reported as the number of seconds required to complete each part, with higher scores reflecting higher degrees of impairment (range 0 - 300 seconds per trial). Normative data are available in the form of demographically adjusted T-scores. The task takes approximately 5 minutes to complete. Clinical trials have repeatedly shown the TMT to be sensitive to the impact of cancer and treatment-related neurotoxicities. Breast cancer survivors have been shown to produce z-scores of 0.56 ± 1.29 on part A and 0.15 ± 1.22 on part B.
Cognitive Function other than working memory (CIFA) | Before and after study intervention on Days 1-5
  The measurement tools for objective cognitive function for this objective will be the Calibrated Ideational Fluency Assessment (CIFA). The CIFA verbal fluency trials are designed to evaluate verbal fluency and executive functioning. The task requires patients to name as many words as possible beginning with two different letters (letter fluency) and that belong to two different categories (category fluency) over four separate one-minute trials. The task takes approximately five minutes to complete. Scoring is based on the number of correct words produced over the course of the four trials, with greater values reflecting better performance. Normative data are available in the form of demographically adjusted T-scores.
Chemotherapy administration | End of study (approximately 3 weeks)
  Chemotherapy will be considered to be given on time if there is no more than 3 days delay (i.e. administered within 24 days of prior cycle of docetaxel-based chemotherapy). Timeliness of administration of chemotherapy after tDCS will be evaluated by chart review to determine if the next cycle of docetaxel-based chemotherapy is administered within 24 days of the chemotherapy administered during study participation and prior to tDCS (i.e. no more than 3 day delay in a 21 day cycle). This endpoint will only be evaluated in participants for whom an additional cycle of docetaxel-based chemotherapy is planned.
Medical Record Review | Baseline and End of study (approximately 3 weeks)
  Available medical records will be reviewed in the electronic medical record to obtain information relative to factors which may impact the feasibility of tDCS and the effect of tDCS on fatigue, cognitive function and quality of life. Information obtained from charts may include but will not be limited to: breast cancer stage, baseline hemoglobin, # of prior cycles of docetaxel-based chemotherapy, concurrent cancer therapy, prior breast cancer surgery, prior breast cancer radiation, prior breast cancer systemic therapy, hormone receptor status, HER2 status, concurrent medications at study enrollment, substance use history, mental health history, marital status, history of thyroid disease, history of cerebrovascular disease, family history of neurologic disease, history of cardiopulmonary disease, steroid dose prior to docetaxel administration, supportive care medications and any other comorbid medical conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Smith, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
For the feasibility endpoint, we will report the count, proportion, and 90% confidence interval of participants completing at least 4 tDCS sessions. The summary statistics will be reported by study arm and for all patients.